CLINICAL TRIAL: NCT00983879
Title: A Longitudinal Observational Study That Will Evaluate Prospectively Clinical and Surrogate Parameters That Are Affected in Infant Patients With Globoid Cell Leukodystrophy
Brief Title: The Natural History of Infantile Globoid Cell Leukodystrophy
Status: Completed | Type: Observational
Sponsor: Zymenex A/S (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: rhGALC-01
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Infantile Globoid Cell Leukodystrophy
Keywords: Infantile globoid cell leukodystrophy; GLD; Krabbe disease; Natural History Study
MeSH Terms: conditions — Leukodystrophy, Globoid Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this natural history study is to understand more about the progression of infantile Krabbe disease, a very rare genetic disease. There is very little published longitudinal data with only anecdotal cases. This natural history study will be important in understanding the effect of future therapies that are presently in the preclinical phase.

DETAILED DESCRIPTION:
Infantile globoid cell leukodystrophy (GLD, or Krabbe disease) is a rare, inherited degenerative disorder of the central and peripheral nervous systems. It is characterized by the presence of globoid cells (multinucleated cells), the breakdown of the nerve's protective myelin coating, and destruction of brain cells. Globoid cell leukodystrophy is one of a group of genetic disorders called the leukodystrophies. These disorders impair the growth or development of the myelin sheath, and causes severe degeneration of mental and motor skills. Myelin, which lends its color to the "white matter" of the brain, is a complex substance made up of a number of different glucoproteins and glucolipids, the most important of which is galactocerebroside. Each of the leukodystrophies affects one of these substances. Globoid cell leukodystrophy is caused by a deficiency of galactocerebroside ß-galactosidase (GALC), an essential enzyme for myelin metabolism. The disease most often affects infants, with onset before the age of 6 months, but can occur in adolescence or adulthood. Symptoms include irritability, unexplained fever, limb stiffness (hypertonia), seizures, feeding difficulties, vomiting, and slowing of mental and motor development. Other symptoms include muscle weakness, spasticity, deafness, and blindness.

There is no cure for globoid cell leukodystrophy. Generally, treatment for the disorder is symptomatic and supportive.

Infantile globoid cell leukodystrophy is generally fatal before age 2 years. Patients with juvenile- or adult-onset disease generally have a milder course of the disease and live significantly longer.

Globoid cell leukodystrophy is a autosomal recessive disorder with a wide geographic distribution. The incidence in the United States is estimated as 1 in 100.000 births. However, the incidence appears to be higher in the Scandinavian countries. 32 Swedish cases were reported during the period from 1953 through 1967 with calculated incidence at 1.9 per 100.000 births.

To be able to compare the benefits experienced by infants with globoid cell leukodystrophy, who receive a possible future treatment, to those untreated, a better understanding of the natural course of infantile GLD is necessary. The current literature contains only case studies of individual or small groups of GLD patients. A longitudinal study of a larger population of patients with infantile GLD has yet to be performed. This protocol is a 1.5 years longitudinal observational study to capture natural history data in patients with infantile GLD. This data will provide information on the range and diversity of clinical disease parameters that can in the future be used to evaluate treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. (Study-related activities are any procedure that would not have been performed during normal management of the subject)
* The patient must have a documented diagnosis of infantile globoid cell leukodystrophy with galactocerebroside ß-galactosidase (GALC) activity < 0.50 nmol/h/mg protein and evidence of two pathogenic mutations in the GALC gene must be confirmed after the baseline visit
* The patient must have an age at the time of screening < 2 years
* The patient's parent(s) and/or legal guardian must have the ability to comply with the clinical protocol

Exclusion Criteria:

* History of hematopoietic stem cell transplantation
* Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition
* Presence of major congenital abnormality
* Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the principal investigator, would preclude participation in the study
* Use of any investigational product within 30 days prior to study enrollment or currently enrolled in another study which involves clinical investigations
* The patient's parent(s) and/or legal guardian is unable to understand the nature, scope, and possible consequences of the study
* Patient is unable to comply with the protocol, i.e. inability to return for follow-up evaluations or otherwise unlikely to complete the study as determined by the principal investigator

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will be enrolled regardless of gender, race or ethnicity. Patients will be identified through clinical referrals from other physicians or medical centers and also those patients receiving clinical care at the Program for Neurodevelopmental Function in Rare Disorders.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
This longitudinal observational study will collect information on patients diagnosed with infantile globoid cell leukodystrophy over approximately an 18-month period. | 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Escolar, MD, Principal Investigator — NFRD Office, Pittsburgh, Pennsylvania, US
Locations (1):
- Children's Hospital of Pittsburgh, 4401 One Children's Hospital Drive,4401 Penn Avenue, Pittsburgh, Pennsylvania, United States